CLINICAL TRIAL: NCT03228693
Title: Gene Expression and Biomarker Profiling of Keloid Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Roopal Kundu, Associate Professor of Dermatology and Medical Education, Northwestern University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RVK 09062016
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Keloid; Keloid of Ear Lobe; Healthy Adults
Keywords: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Active Comparator): Baseline lesional and non-lesional biopsies and re-biopsy 6-8 weeks later with intralesional triamcinolone injections at 9-10, 12-16, and 24-32 weeks.
  Interventions: Procedure: Biopsy and/or triamcinolone injection
- Group 2 (Active Comparator): Baseline lesional biopsy and re-biopsy at 6-8 weeks with intralesional triamcinolone injections at 3-4, 9-10, 12-16, and 24-32 weeks
  Interventions: Procedure: Biopsy and/or triamcinolone injection
- Group 3 (Active Comparator): Baseline lesional and non-lesional biopsy and re-biopsy 3-4 months later with intralesional triamcinolone injections at 18-20 and 24-32 weeks.
  Interventions: Procedure: Biopsy and/or triamcinolone injection
- Group 4 (Active Comparator): Baseline lesional biopsy and re-biopsy at 3-4 months with intralesional triamcinolone injections at 3-4, 6-8, 18-20 and 24-32 weeks.
  Interventions: Procedure: Biopsy and/or triamcinolone injection
- Group 5 (Active Comparator): Normal patient skin (surgical or adjacent to other biopsy) from subjects with no self-reported history of keloids.
  Interventions: Procedure: Biopsy and/or triamcinolone injection
- Earlobe Keloid (Other): Complete excision of an earlobe keloid measuring > 10mm will be taken.
  Interventions: Procedure: Excisional Biopsy

INTERVENTIONS:
Procedure: Biopsy and/or triamcinolone injection — Subjects will have their blood drawn during the first study visit. Subsequently, a punch biopsy and/or triamcinolone injection will be given based on group timeline.
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5
Procedure: Excisional Biopsy — Complete excision of an earlobe keloid will be taken.
  Arms: Earlobe Keloid

SUMMARY:
This study aims to examine both the genetic profile and the biomarkers implicated in keloid scar formation.

Hypothesis:

1. Differences in the genetic profiles of lesional and non-lesional skin contribute a given population's propensity to develop keloids
2. Differences in biomolecules expressed in subjects with and without keloids can help predict keloid occurrence and severity
3. Biomarker analysis will provide useful insights for future targeted therapies for keloid scars

DETAILED DESCRIPTION:
Objectives:

1. Determine gene expression profiles of keloid scar tissue using samples collected longitudinally
2. Define and compare the molecular biomarkers of keloid scars in keloid (lesional) and non-lesional skin biopsies and serum samples from adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Patient with an untreated keloid scar or a patient with a keloid scar that has not had treatment for at least 6 months before time of enrollment
* Patients without keloids coming into the dermatology clinic for a keloid unrelated issue (Group 5 only)

Exclusion Criteria:

* Patients who have had treatment of their keloid scar within 6 months of date of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Keloid progression | One year
  Assess effectiveness of triamcinolone injection (keloid size measured in millimeters)
Gene Expression | One year
  Blood will be drawn during first study visit for analysis
Keloid recurrence | One year
  Assess keloid recurrence at biopsy site (measured by number of keloids)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Kundu, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided